CLINICAL TRIAL: NCT05978154
Title: Thigh Muscle Mass and Muscle Wasting in Patients in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Ansan Hospital (Other)
Responsible Party: Principal Investigator, Ahn, Sejoong, Korea University Ansan Hospital, Korea University Ansan Hospital
Other Study IDs: musclemassandwastingined
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Sepsis; Cardiac Arrest; Acute Respiratory Failure; Patients Who Visit Emergency Department; Shock; Trauma
MeSH Terms: conditions — Sepsis; Heart Arrest; Shock; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Thigh muscle mass and muscle wasting (exposure) — Thigh muscle mass and muscle wasting (exposure variable)

SUMMARY:
The goal of this observational study is to evaluate whether thigh muscle mass and muscle wasting are associated with mortality in patients who visit the emergency department. The main questions it aims to answer are:

* Is thigh muscle mass associated with mortality in patient who visit the emergency department?
* Does muscle wasting exist during staying in the emergency department?
* Is muscle wasting associated with mortality in patient who visit the emergency department? Participants will be evaluated for serial thigh muscle mass using point-of-care ultrasound at the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* patients who visit the emergency department of Korea University Ansan Hospital during study period
* patients with age within the limits
* patients who are willing to be participate the study with informed consent
* patients who undergo point-of-care ultrasound to evaluate thigh muscle mass

Exclusion Criteria:

* patients with age out of limits
* patients who have deformities on lower leg
* patients who is unable to maintain appropriate position to undergo point-of-care ultrasound
* patients who decline to participate the study
* patients who have 'do-not-resuscitate' order or are not willing to be resuscitated
* patients of whom point-of-care ultrasound on thigh muscle mass was not performed

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who visit the emergency department with informed consent and then who undergo point-of-care ultrasound to evaluate thigh muscle mass.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
28 day mortality | 28 days after study enrollment
  28 day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Ansan Hospital, Ansan-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No